CLINICAL TRIAL: NCT03471676
Title: Study of the Correlation Between Muscle Oxygenation and Motor Function in Children With Neuromuscular Disease.
Acronym: OXMNM
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI17/OXMNM; 2017-A02931-52 (Other: IdRCB); 17.11.07 (Other: CPP)
Record Dates: First submitted 2018-03-02; First posted 2018-03-20 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Neuromuscular Diseases in Infants; Neuromuscular Diseases in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Muscular oximetry: 6 minutes walking test performed in the routine medical care with muscle oximetry recording in children suffering from neuromuscular diseases
  Interventions: Other: Muscular oximetry

INTERVENTIONS:
Other: Muscular oximetry — 6 minutes walking test performed in the routine medical care with muscle oximetry recording

SUMMARY:
Preliminary data underline the fact that muscular deoxygenation during training happens earlier in adult patients suffering from neuromuscular disorders in comparison to controls. Up to date, pediatric data are lacking.

The study aims at demonstrating if a correlation exists between the motor deficiency and the muscular deoxygenation in children suffering from neuromuscular disorders.

DETAILED DESCRIPTION:
Preliminary data underline the fact that muscular deoxygenation during training happens earlier in adult patients suffering from neuromuscular disorders in comparison to controls, as it was demonstrated in Becker muscular dystrophy patients and fascioscapulo humeral muscular dystrophy. Moreover, the deoxygenation kinetics was positively correlated to the functional status and the muscular deficiency severity. However, no pediatric study has been conducted on this topic up to date.

The aim of the study is to determine if a correlation exists in children suffering from neuromuscular diseases:

* between muscular oxygenation and the percentage of the 6 minutes walking test performed in the routine medical care
* between muscular oxygenation and the total and D1 motor function measure value

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 18 years-old suffering from a neuromuscular disorder
* Able to walk, with or without help

Exclusion Criteria:

* Hypoxia secondary to heart or lung disease
* Visual impairment (<5/10)
* Parents refusal concerning data storage

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 6-17 years old patients suffering from neuromuscular disorder and able to walk
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Muscular oxygenation | 6 minutes
  Muscular oximetry

SECONDARY OUTCOMES:
6 minutes walking distance | 6 minutes
  6 minutes walking distance
Motor function | 25 minutes
  Motor function measure (MFM scale)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle LAGRUE, MD, PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- University Hospital, Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No